CLINICAL TRIAL: NCT06441318
Title: A Phase 1, Randomized, Partially Double-Blind, Placebo- and Positive-Controlled, Parallel Study to Evaluate the Effect of Povorcitinib on the QT/QTc Interval in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Povorcitinib on the QT/QTc Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB54707-107
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy Participants
Keywords: INCB054707
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Group 1 (Experimental): Povorcitinib and placebo will be administered at the protocol defined doses.
  Interventions: Drug: Povorcitinib; Drug: Placebo
- Treatment Group 2 (Experimental): Povorcitinib will be administered at the protocol defined doses.
  Interventions: Drug: Povorcitinib
- Treatment Group 3 (Placebo Comparator): Placebo will be administered at the protocol defined doses.
  Interventions: Drug: Placebo
- Treatment Group 4 (Active Comparator): Moxifloxacin will be administered at the protocol defined doses.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Povorcitinib — Povorcitinib will be administered at protocol defined dose.
  Other Names: INCB054707
  Arms: Treatment Group 1; Treatment Group 2
Drug: Placebo — Placebo will be administered at protocol defined dose.
  Arms: Treatment Group 1; Treatment Group 3
Drug: Moxifloxacin — Moxifloxacin will be administered at protocol defined dose.
  Arms: Treatment Group 4

SUMMARY:
The purpose of this study is to evaluate the effect of povorcitinib on the QT/QTc Interval in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Age 18 to 55 years inclusive at the time of signing the ICF.
* Body mass index between 18.0 and 30.5 kg/m2, inclusive.
* No clinically significant findings on screening evaluations as determined by the investigator (clinical, laboratory, and ECG).
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening. Participants with any history of myasthenia gravis will be excluded.
* Presence or history of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn disease or chronic pancreatitis).
* Current or recent (within 3 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy and excluding appendectomy and hernia repair) that could affect the absorption of study drug or moxifloxacin.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg at screening, confirmed by repeat testing).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* History of tobacco- or nicotine-containing product-use within 1 month before screening.
* Pregnant or breastfeeding.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in QT interval corrected using Fridericia's formula (QTcF) | Up to Day 3
  Electrocardiogram measurement of the maximum absolute change from baseline in Fridericia's correction for QT interval (QTcF)
Change from Baseline in heart rate (HR) | Up to Day 3
  Electrocardiogram measurement of change from baseline in HR.
Change from Baseline in the PR Interval (PR) | Up to Day 3
  Electrocardiogram measurement of change from baseline in PR.
Change from Baseline in the QRS interval (QRS) | Up to Day 3
  Electrocardiogram measurement of change from baseline in QRS.

SECONDARY OUTCOMES:
Safety and tolerability as measured by the frequency, duration, and severity of adverse events (AEs) | Up to Day 22
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a subject provides informed consent.
Povorcitinib concentration in plasma | Up to Day 7
  Povorcitinib concentration in plasma.
Moxifloxacin concentration in plasma | Up to Day 7
  Moxifloxacin concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion Clinical Research Unit, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No